CLINICAL TRIAL: NCT00678626
Title: A Randomized Phase 2, Open-Label Study Of CP-751,871 In Combination With Docetaxel And Docetaxel Alone As A First Line Treatment Of Patients With Advanced Breast Cancer
Brief Title: Phase 2 Trial Of CP-751,871 And Docetaxel In Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4021008
Record Dates: First submitted 2008-05-12; First posted 2008-05-15 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: Key words: Docetaxel; breast cancer; breast diseases; breast neoplasms; antineoplastic agents; neoplasms;HER-2 negative; Stage IIIB or IV breast cancer.
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — figitumumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): combination of CP-751,871 + docetaxel administered
  Interventions: Drug: CP-751,871
- Arm B (Active Comparator): chemotherapy
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: CP-751,871 — Docetaxel administered every 3 weeks. CP-751,871 administered every 3 weeks. CP-751,871 administration (20 mg/kg IV) will continue after the docetaxel is stopped.
  Arms: Arm A
Drug: Docetaxel — Docetaxel only is administered every 3 weeks. After progression, administration with CP-751, 871 (20 mg/kg IV) is permitted.
  Arms: Arm B

SUMMARY:
This study will assess the effectiveness of CP- 751,871 when given in combination with docetaxel to women with the first occurrence of advanced breast cancer disease. The effectiveness will be measured by progression-free survival duration. Patients will be followed for 2 years from the date of randomization.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed diagnosis with evidence of either metastatic disease (Stage IV) of locally recurrent disease not amenable to curative resection or radiation therapy (Stage IIIB).
* Her-2negative breast cancer or unknown Her-2 status.
* at least 1 measurable lesion as defined by RECIST.
* ECOG status 0-1
* adequate bone marrow, hepatic and renal function.
* left ventricular ejection fraction of greater than or equal to 50%.
* willingness to discontinue hormonal therapy.

Exclusion Criteria:

* any previous chemotherapy for advanced disease.
* prior exposure to taxanes as (neo) adjuvant treatment less than 12 months prior to randomization.
* symptomatic brain metastases.
* prior anti-IGF-1R based investigational therapy.
* peripheral neuropathy greater than grade 2.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 3 years

SECONDARY OUTCOMES:
Biomarkers (IGF-1R positive Circulating Tumor Cells; Anti-Drug Antibodies) | 3 years
Overall Response | 3 years
Overall Survival | 3 years
Safety and tolerability | 3 years
Patient Reported Outcomes using the MDASI (MD Anderson Symptom Inventory) questionnaire | 3 years
Pharmacokinetics of CP-751,871 | 3 years
Optional tissue markers of the IGF-1R pathway from tumor tissue obtained | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021008&StudyName=Phase%202%20Trial%20Of%20CP-751%2C871%20And%20Docetaxel%20In%20Advanced%20Breast%20Cancer